CLINICAL TRIAL: NCT05044221
Title: Supporting the Recovery Needs of Patients Following Intensive Care
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Melbourne (Other)
Responsible Party: Principal Investigator, Selina M Parry, Cardiorespiratory Team Lead, Department of Physiotherapy, University of Melbourne
Other Study IDs: 2020.333; RMH69389 (Other: ERM)
Record Dates: First submitted 2021-08-30; First posted 2021-09-14 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Post Intensive Care Unit Syndrome; Post Intensive Care Syndrome; ICU Acquired Weakness; Intensive Care Unit Syndrome; Intensive Care Unit Acquired Weakness
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interviews: Past ICU patients and caregivers: Former ICU patients and their families that meet the following criteria: Adults > 18 years and above who required at least 48 hours of invasive mechanical ventilation and were in the ICU at least 4 days with an ICU admission in the past five years; and able to participate in a workshop in English.
  Interventions: Other: Former ICU patient and caregiver workshops
- Interviews: Health care professionals: Active working health professionals with prior experience working directly in the ICU setting and/or care for ICU patients in their own clinical rea (acute, subacute and/or community settings).
  Interventions: Other: Health care professional workshops

INTERVENTIONS:
Other: Former ICU patient and caregiver workshops — In depth interviews and workshops will be conducted with individuals enrolled in the study.
  Other Names: In depth interviews and workshops
  Groups: Interviews: Past ICU patients and caregivers
Other: Health care professional workshops — In depth interviews and workshops will be conducted with individuals enrolled in the study.
  Other Names: In depth interviews and workshops
  Groups: Interviews: Health care professionals

SUMMARY:
Recovery for intensive care survivors is limited by ongoing problems with walking, strength, fatigue, mental distress and cognitive morbidity known as 'Post Intensive Care Syndrome'. There has been increasing interest in ways that clinicians can support patients in their post ICU recovery.

The investigators are undertaking a co design approach to informing the design of a recovery pathway for patients who have been admitted to the intensive care to support them in their return to home, family and working responsibilities.

DETAILED DESCRIPTION:
This project will aim to involve ~ 20 past ICU patient/family members and ~20 health professionals to participate in a co-design approach to examine the recovery needs and resources that are required to support patients after leaving hospital. Using an experience based co design methodology three 2-hour workshops will be run with the first workshop involving patients/family members, the second involving healthcare professionals to separately gain thoughts and perspectives, and then the final workshop which will be combined to identify and problem solve priority resources and solutions.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized adults, aged 18 years or over
* Admitted to the ICU requiring invasive mechanical ventilation for > 48 hours and remain in the ICU for a minimum of four days
* Living at home before the current admission (not in a facility and/or no fixed abode)

Exclusion Criteria:

* Non-English speaking (insufficient English language skills to read and understand questionnaires and patient information consent form)
* Pre-existing documented cognitive impairment
* Spinal cord injury or other primary neuromuscular disease
* New lower limb fracture with altered weight bearing status
* Expected survival < 3 months according to the treating medical team
* Active substance abuse or psychosis
* Lack of access to telephone / computer or inability to use these resources independently (which would impact on ability to complete the intervention)
* Pregnancy
* Suicidality
* Incarcerated
* Cardiac surgery within this ICU admission (as these patients routinely receive a standard outpatient rehabilitation through cardiac rehabilitation)
* Poor premorbid mobility defined as < 10 metres ambulation +/- gait aid independently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited across two Australian hospitals
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Lived experiences and opinions | 3 months
  Capability Opportunity Motivation Barriers and Theoretical Domains Framework will be used to interpret qualitative data from the workshops and interviews.

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - The Royal Melbourne Hospital, Melbourne, Victoria
  - St Vincent's Hospital Melbourne, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] da Silva AA, Granger CL, Abo S, Sheehan J, Barson E, Beach L, Pound G, Ali Abdelhamid Y, Fetterplace K, Fini NA, Merolli M, Sloan E, Parry SM. "How Do I Test the Waters? How Do I Go Forward?": Codesigning a Supportive Pathway after Critical Illness. Ann Am Thorac Soc. 2024 Jun;21(6):916-927. doi: 10.1513/AnnalsATS.202307-599OC. PMID 38330169